CLINICAL TRIAL: NCT04330521
Title: Impact of the Coronavirus (COVID-19) on Patients With Cancer
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Manali Indravadan Patel, Assistant Professor, Stanford University
Other Study IDs: 55596
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Cancer; COVID-19
Keywords: Coronavirus; COVID-19; Cancer; Life Change Events
MeSH Terms: conditions — Neoplasms; COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to understand the impact of COVID-19 on patients with cancer through a survey.

DETAILED DESCRIPTION:
The global spread of coronavirus (COVID-19) is affecting cancer patients and their treatments. Cancer patients are among those at high risk of developing serious illness from an infection because their immune systems are often weakened by cancer and its treatments. Due to the growing coronavirus outbreak, patients clinic visits are being cancelled and many are facing social isolation and strict restrictions on their daily lives. We want to evaluate the impact of the coronavirus on the patient's well-being and their cancer care by assessing the delays in their medical care and any other unmet needs. We have created a survey that is available online for any patient with cancer to fill out voluntarily regarding their experiences to date. The survey is available at: https://stanforduniversity.qualtrics.com/jfe/form/SV_ctKS6ZSMYdEYoXX

ELIGIBILITY:
Inclusion Criteria:

1. The patients must be 18 years or older.
2. Patients who opt in to complete the survey.
3. Patients must have the capacity to verbally consent for the interview.

Exclusion Criteria:

1.Patients who under the age of 18 years old.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who are diagnosed with any cancer diagnosis . We plan to enroll as many patients as possible in the survey portion of the study - we have no limitation of the numbers and do not require a specific number to participate although we hope to achieve at least 50 participants who fill out the survey.
  Among survey participants, we plan to enroll 18-30 participants in semi-structured telephone interviews. These participants will be randomly selected among those who filled out the survey.
  The research procedures are as followed:
  1. Survey: An online survey link will include questions regarding the impact patients with cancer are experiencing during the coronavirus outbreak.
  2. Semi-structured Interviews (18-30 participants): For those participants who state that they would like to participate in an interview, a random sample will be contacted.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-04-08 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants who fill out the survey and participate in the semi-structured interviews. | 12 Months
  We will track the number of participants who fill out the survey for the 12 month duration of the study and the number of participants who participate in the semi-structured telephone interviews.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Impact of the novel Coronavirus (COVID-19) on Patients with Cancer Qualtrics Survey — https://stanforduniversity.qualtrics.com/jfe/form/SV_ctKS6ZSMYdEYoXX